CLINICAL TRIAL: NCT02664285
Title: Closure Versus Non Closure of Subcutaneous Tissue After Cesarean Section in Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rehab Mohamed Abdelrahman, Lecturer of Obstetrics and Gynaecology Faculty of Medicine, Ain Shams University, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ceserean section
Record Dates: First submitted 2016-01-20; First posted 2016-01-27 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Abdominal Delivery

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- closure of subcutaneous tissue (Other): in diabetic patients, the subcutaneous fat will be closed with three to five interrupted sutures. The sutures were tied until the tissue was adequately re-approximated, but not as hard as possible to avoid necrosis after cesarean section.
  Interventions: Other: closure of subcutaneous tissue
- No closure of subcutaneous tissue (Other): in diabetic patients, the subcutaneous fat will not sutured after cesarean section.
  Interventions: Other: No closure of subcutaneous tissue

INTERVENTIONS:
Other: closure of subcutaneous tissue — the subcutaneous fat will be closed with three to five interrupted sutures. The sutures were tied until the tissue was adequately re-approximated, but not as hard as possible to avoid necrosis after cesarean section in diabetic patients.
  Arms: closure of subcutaneous tissue
Other: No closure of subcutaneous tissue — the subcutaneous fat will not sutured after cesarean section in diabetic patients.
  Arms: No closure of subcutaneous tissue

SUMMARY:
The aim of this study is to determine the surgical site infection rate and the patient's satisfaction for closure of subcutaneous tissue versus non closure of subcutaneous tissue after cesarean delivery in women with diabetes mellitus.

DETAILED DESCRIPTION:
This is a randomized prospective comparative clinical study will be conducted in Ain Shams University, Maternity Hospital.

This study will include a sample of (136) pregnant women with gestational diabetes mellitus and type 2 diabetes mellitus who underwent elective Cesarean section.

Patients will b divided into two groups:

Group A (closure group): will include 68 pregnant women who underwent elective Cesarean section with closure of subcutaneous tissue. Group B (non closure group): will include 68 pregnant women who underwent elective Cesarean section without closure of subcutaneous tissue.

• All participants in the study will have consent.

All included women will be subjected to the following:

1. History Full history taking, (personal, present, past and obstetrics history).
2. Clinical examination including:

General examination:

1. Assessment of vital data
2. Assessment of general condition.
3. Cardiac and chest examination, to exclude any contraindication for anesthesia.

Abdominal examination:

Assessment of fundal level for fetal dating, fetal lie and fetal heart sound. 3. Investigations: Laboratory Complete blood picture.- Random blood sugar.

Ultrasonography:

Fetal biometry for fetal dating and fetal viability. 4. All participants operated under general or spinal anesthesia. Prophylactic antibiotic is given according to the approved protocol of Ain Shams Maternity Hospital (as two intravenous doses of broad spectrum penicillin (after clamping of the umbilical cord and 12 hours postoperatively. Oral antibiotic of the same group was then started for 3-5 days.

5.In group A (closure group)the subcutaneous fat will be closed with three to five interrupted sutures. The sutures were tied until the tissue was adequately re-approximated, but not as hard as possible to avoid necrosis. In group B (non closure group) the subcutaneous fat will not sutured.

6.In all participants Skin to be closed by subcuticular stitches using absorbable polyglactin 910 suture 7. Dressing is removed after 48hours postoperatively, to be disinfected with alcohol 70% antiseptic solution daily in both groups.

8. The wound is to be inspected 48 hours, 7 days and one month after the cesarean section.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women in childbearing period (18-45 years).
2. Women planned for elective cesarean section.
3. Pregnant women with gestational diabetes according to medical records.

Exclusion Criteria:

1. Hemoglobin less than 10g/dl.
2. Intra operative events that may themselves predispose to postoperative infection (e.g. operative time more than 90 minutes).
3. Rupture of membrane more than 12 hours.
4. Receive corticosteroid medications.
5. Immunosuppressive disease or Auto immune disease.
6. Concurrent infection (e.g. signs of pyelonephritis, chest infection).
7. Previous history of two C.S.
8. Previous laparotomy other than C.S.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2016-01; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with surgical site infection | 9 months
  Surgical site infection: including the following manifestations: Collection; inflammatory signs (pain, tenderness, edema, redness); dehiscence (wound separation) or positive culture.

SECONDARY OUTCOMES:
Number of participants with wound seroma | month
  wound seroma, superficial wound breakdown (defined as skin and/or subcutaneous dehiscence with intact fascial layer).
Number of participants with postoperative pain | 24 hours
  Postoperative pain (judged after 24 hours, through visual analogue scale (VAS); with 0 meaning no pain, and 10 meaning the worst pain).
Number of participants with postoperative fever | 48 hours
  postoperative fever (defined as temperature more than thirty eight degree, 48 hours postoperative.
Number of participants with cosmetic wound | 1 month
  Is cosmetic wound outcome for one month postoperative good or no?

IPD SHARING:
Plan to Share IPD: Yes
The aim of this study is to determine the surgical site infection rate and the patient's satisfaction for closure of subcutaneous tissue versus non closure of subcutaneous tissue after cesarean delivery in women with diabetes mellitus.